CLINICAL TRIAL: NCT00429325
Title: Comparative Evaluation of Accuracy of Fecal Calprotectin, Lactoferrin and Occult Blood Testing (FOBT) in Predicting Microbiological Diagnosis for Acute Infectious Diarrhea: A Prospective Multicentre Double Blind Randomized Controlled Trial.
Brief Title: Fecal Calprotectin: Cheap Marker for Diagnosing Acute Infectious Diarrhea
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: JWGUH-2
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-02

CONDITIONS: Acute Diarrhea
Keywords: acute infectious diarrhea,; fecal calprotectin,; stool culture,; hemoccult test,; Guaiac fecal occult blood test (FOBT); fecal lactoferrin

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Every year more than 4 billion cases of diarrhea occur worldwide culminating in about 2.5 million deaths, almost all in the developing nations. Reliable diagnosis of patients with acute infectious diarrhea which could be appropriately managed with antibiotics at presentation still remains a formidable challenge to the clinicians. To address this issue of predicting microbiological infectious etiology for diagnosing acute infectious diarrhea, we would evaluate stools from all patients with acute diarrhea with culture, Guaiac based fecal occult blood test (FOBT), Calprotectin and lactoferrin assays simultaneously. This would be the first study evaluating fecal calprotectin as a diagnostic marker in acute diarrhea

DETAILED DESCRIPTION:
There are about 4 billion cases of diarrhea worldwide i.e. about half the population of the world is affected with it once every year. Though the mortality because of it has reduced significantly still it contributes to more than 2.2 million deaths (4% of all deaths) and 5% of health loss due to disability annually. Most of these deaths are due to acute diarrhea, in the developing countries which rapidly causes dehydration unless adequately supplemented. Unlike many of the medical challenges, acute infectious diarrhea still remains a significant global health hazard. Adequate, appropriate treatment with proper antimicrobials not only shortens the morbidity, hospitalisation and costs to the society but also can be life saving in certain infectious diarrhea.

The biggest problem is the lack of accurate diagnostic modality to differentiate acute infections from non infectious diarrhea. Stool microscopy, Guaiac based fecal blood tests (hemoccult), lactoferrin assays and bacteriological culture have been used for this purpose till now. However none of these were of great help in the diagnostic algorithm of management of acute diarrhea. The gold standard to diagnose acute infectious diarrhea is of course the bacteriological culture. But its very expensive, time consuming and delays definite therapy. There is a need for something simple, cheap, fast and accurate to diagnose acute infectious diarrhea. In the present prospective study, we plan to evaluate the performance characteristics of fecal calprotectin in diverse group of patients referred to our hospitals. Its performance characteristics would be compared with that of lactoferrin and FOBT.

ELIGIBILITY:
Inclusion Criteria:

* All patients having acute diarrhea i.e. 3 or more stools per day or stool weight exceeding 200 grams lasting less than 15 days

Exclusion Criteria:

Patients having the following diagnosis as they might have high calprotectin levels not only because of the diarrhea per se but may also be because of the underlying pathology itself.

* Inflammatory bowel disease (Crohn's disease, ulcerative disease)
* Gastrointestinal malignancy (colorectal cancer, gastric cancer etc)
* Cirrhosis of liver
* Chronic pancreatitis
* Currently on non steroidal anti inflammatory therapy
* Younger than 1 year of age

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2004-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen M Stein, MD,PhD, Study Director — JW Goethe University Hospital, Frankfurt; Yogesh M Shastri, MD, DNB, Principal Investigator — JW Goethe University Hospital, Frankfurt; Wolfgang F Caspary, MD, Study Chair — JW Goethe University Hospital, Frankfurt
Locations (2):
- Germany (2):
  - Laboratory Walther, Weindel & Colleagues, Frankfurt am Main, Hesse
  - Department of Medicine I, Division of Gastroenterology and Clinical Nutrition, Johann Wolfgang Goethe-University Hospital, Frankfurt am Main, Hesse